CLINICAL TRIAL: NCT04440202
Title: Cardioprotective Properties of Sea Bream Bred With a Fraction of Polar Lipids Extracted From Olive Oil By-products: the ELAIOTSIPOURA Study
Brief Title: Cardioprotective Properties of ELAIOTSIPOURA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Collaborators: Nireus Aquaculture (Unknown); University of Thessaly (Other); Cretan Herbalchem S.A. (Unknown); National and Kapodistrian University of Athens (Other); European Regional Development Fund (project code: T1EDK- 00687) (Unknown)
Responsible Party: Principal Investigator, Smaragdi Antonopoulou, Professor in Biochemistry, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71777/13-2-2018
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2022-01

CONDITIONS: Cardiometabolic Health
Keywords: fish; sea bream; dietary intervention; olive oil; polar lipids; platelet aggregation; thrombosis; inflammation; cardioprotection
MeSH Terms: conditions — Thrombosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional sea bream group (Active Comparator): This arm will consume 2 portions (each 200 g cooked) of conventional fish (sea bream) fillet per week for a 1-month period.
  Interventions: Behavioral: Conventional sea bream
- Enriched sea bream group (Experimental): This arm will consume 2 portions (each 200 g cooked) of fish fillet bred with bioactive lipids from olive oil by-products per week for a 1-month period.
  Interventions: Behavioral: Enriched sea bream

INTERVENTIONS:
Behavioral: Conventional sea bream — Participants initially randomized to this intervention arm will be provided with a total of 8 conventional sea bream fillets and will be asked to consume them twice weekly for 1 month. Conventional sea bream fillets will be produced by a fish farming company using standard procedures. Participants will also be instructed to keep the reception of prescribed medications and dietary supplements stable and not to change their lifestyle habits (e.g. other dietary habits besides fish consumption, physical activity habits or sleep habits) during the intervention. After a 1-month wash-out period (no fish consumption), participants will cross over to the other intervention arm.
  Arms: Conventional sea bream group
Behavioral: Enriched sea bream — Participants initially randomized to this intervention arm will be provided with a total of 8 enriched sea bream fillets and will be asked to consume them twice weekly for 1 month. Enriched sea bream fillets will be produced by a fish farming company from fish bread with a diet enriched with a fraction of bioactive polar lipids extracted from olive oil by-products. Participants will also be instructed to keep the reception of prescribed medications and dietary supplements stable and not to change their lifestyle habits (e.g. other dietary habits besides fish consumption, physical activity habits or sleep habits) during the intervention. After a 1-month wash-out period (no fish consumption), participants will cross over to the other intervention arm.
  Arms: Enriched sea bream group

SUMMARY:
Several studies over the last decades have demonstrated the important role of nutrition for either the prevention of chronic diseases, such as cardiovascular disease and cancer, or the increase of their risk. One dietary component with several health benefits as supported by several epidemiological and clinical studies is fish consumption. Both the European Society of Cardiology and the American Heart Association recommend the consumption of at least two servings of fish per week for protection against cardiovascular disease. Nevertheless, the growth of the human population and the rising consumers' awareness, result in a constantly increasing demand for the supply of fish. Aquaculture is significantly contributing to fish supplies all over the world and over the past few years, important breakthroughs have occurred in the replacement of fish oil, traditionally used in aquacultures, by plant oils in compounded fish feeds as a mean to improve the nutritional value of the produced fish. Under this perspective, the utilization of olive oil by-products, widely available in the Mediterranean countries, in fish feeds could result in significant economic and environmental impact. Therefore, the aim of the present double-blind, randomized, crossover clinical trial is to explore the potential cardioprotective properties of "elaiotsipoura", a novel sea bream fed with bioactive lipids isolated from olive oil by-products, against conventionally fed sea bream, in apparently healthy volunteers.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) represent a major public health challenge and the leading cause of mortality worldwide. The elucidation of CVD pathogenesis, as well as the identification of efficient strategies for their prevention and treatment, have been the subject of intense research in recent years. The platelet activation factor (PAF) is one of the most important mediators of atherosclerosis, given that it is produced by cells involved in the formation of atherosclerotic plaque (e.g. endothelial cells, platelets, smooth muscle cells, macrophages and neutrophils) under conditions that predispose to CVD, i.e. inflammation, oxidative stress, endothelial dysfunction and dyslipidaemia. PAF acts on neighbouring cells by inducing a series of responses (e.g. chemotaxis, expression of adhesion molecules and accumulation of platelets) that eventually lead to endothelial and atherosclerotic damage.

The Mediterranean diet (MD) is a dietary pattern with well-established protective effects against the development of CVD. Several foods representative of the MD, such as honey, wine and fish, have been found to be rich in nutrients, mainly of lipid nature, that can act as PAF inhibitors. Investigators have recently focused on olive oil, from which a bioactive polar lipoid (BPL) fraction with strong PAF inhibitors was extracted. The most important of these inhibitors were structurally classified and found to belong to the class of glycolipids. This BPL fraction showed strong anti-atherogenic properties in hypercholesterolaemic rabbits, stronger than those produced by the same amount of olive oil. BPLs could therefore be a bioactive extract that could potentially be used as an additive in biofunctional foods or as a dietary supplement, aiming at preventing atherosclerosis and CVD. However, olive oil cannot be systematically used as the source of such an extract, since the large quantities of olive oil required to extract BPLs combined with its high price make olive oil an unsustainable raw material. In this context, olive oil by-products could be a more suitable alternative source, and their extract has been found to be rich in phenolic compounds and to exert a similar inhibitory effect against PAF. This alternative extract has already been tested in hypercholesterolaemic rabbits and was shown to significantly reduce the thickness of atherosclerotic lesions. In addition, it has already been used by "Nireus Aquaculture" for pilot fish farming.

The aim of the present study is to evaluate the potential cardio-protective properties of an innovative fish bred with bioactive lipids derived from olive oil by-products.

The study will be a randomized, cross-over, double blind clinical trial. The study sample will consist of 30 apparently healthy volunteers aged 35-70 years, with a body mass index of 25-35 kg/m2, who will not be under certain types of medication, namely antidiabetic, anxiolytics/ antidepressants and cortisol. Other prescribed medications and dietary supplements will be allowed, provided that their reception will remain stable by participants throughout the trial. Individuals with diabetes mellitus, active cancer, cardiovascular diseases, chronic inflammatory diseases or psychiatric diseases, as well as those on a weight-loss diet or with recent significant changes in their lifestyle habits will be excluded from the study. Participants will consume 2 servings per week of either a conventional sea bream fillet or an enriched with bioactive lipids derived from olive oil by-products sea bream fillet (serving size: 200 g cooked fish) for 4 weeks, with a 4-week wash-out period between the two interventions. The study physician will be on a weekly contact with each participant to systematically record potential side-effects and will be in charge of terminating the intervention if needed.

Participants will be assessed in terms of lifestyle habits (dietary and physical activity habits), and blood samples will be collected, both at the beginning and end of each intervention period (a total of 4 assessments). Dietary habits will be assessed through a validated for the Greek population food frequency questionnaire, while physical activity level will be assessed through the Athens Physical Activity Questionnaire, also validated in the Greek population. Adherence to dietary intervention will be assessed through weekly self-monitoring diaries, in which participants will record the exact day and quantity of fish they consumed. Participants' diastolic and systolic blood pressure will be measured by the study physician at the 4 assessments throughout the study. All blood samples will be collected and analyzed in the Laboratories of Clinical Nutrition and of Biology, Biochemistry, Physiology and Microbiology of the Department of Nutrition and Dietetics of Harokopio University of Athens by experienced personnel. The ability of the platelet-rich plasma (PRP) to be accumulated under the influence of PAF and adenosine diphosphate (ADP) will be assessed by calculating the corresponding efficiency concentration fifty (EC50) values. A priori statistical power analysis showed that 25 participants in each arm were required to achieve statistical power equal to 83% at 5% significance level of two-sided hypotheses that evaluated 1 standard deviation (SD) differences based on EC50 values of platelet aggregation induced by PAF. In addition, thrombosis markers, oxidation and inflammation markers, as well as glycemic and lipidemic profile parameters, will be measured in participants' blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35-70 years old
2. Body mass index 25-35 kg/m2
3. Habitual fish consumption ≤1 portion/week (1 portion: 150 g cooked fish)

Exclusion Criteria:

1. Presence of diabetes mellitus, active cancer, cardiovascular disease, chronic inflammatory or psychiatric diseases
2. Reception of antidiabetic, anxiolytic, antidepressant or cortisol medication
3. Habitual excessive alcohol intake (>210 g of ethanol/week for men and >140 g of ethanol/week for women)
4. Currently on a weight-loss diet or recent change (within 6 months) in lifestyle habits

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of adenosine diphosphate-induced platelet aggregation at 4 weeks | 0 (baseline) and 4 weeks
  Efficiency concentration fifty of adenosine diphosphate-induced platelet aggregation (microM) will be assessed by light transmittance aggregometry
Change from baseline of platelet activating factor-induced platelet aggregation at 4 weeks | 0 (baseline) and 4 weeks
  Efficiency concentration fifty of platelet activating factor-induced platelet aggregation (microM) will be assessed by light transmittance aggregometry
Change from baseline in tissue plasminogen activator activity at 4 weeks | 0 (baseline) and 4 weeks
  Tissue plasminogen activator activity (mIU/mL) will be measured in blood samples using commercially available ELISA kits
Change from baseline in of plasminogen activator inhibitor-1 activity at 4 weeks | 0 (baseline) and 4 weeks
  Plasminogen activator inhibitor-1 activity (mAU/mL) will be measured in blood samples using commercially available ELISA kits

SECONDARY OUTCOMES:
Change from baseline in high sensitivity interleukin-6 levels at 4 weeks | 0 (baseline) and 4 weeks
  High-sensitivity interleukin-6 levels (pg/mL) will be measured in blood samples using commercially available ELISA kits
Change from baseline in high sensitivity interleukin-10 levels at 4 weeks | 0 (baseline) and 4 weeks
  High-sensitivity interleukin-10 levels (pg/mL) will be measured in blood samples using commercially available ELISA kits
Change from baseline in soluble P-selectin levels at 4 weeks | 0 (baseline) and 4 weeks
  Soluble P-selectin levels (ng/mL) will be measured in blood samples using commercially available ELISA kits

CONTACTS AND LOCATIONS:
Overall Officials: Smaragdi Antonopoulou, PhD, Principal Investigator — Department of Nutrition and Dietetics, Harokopio University; Tzortzis Nomikos, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University; Elizabeth Fragopoulou, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University; Meropi D Kontogianni, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University; Michael Georgoulis, PhD, Study Chair — Department of Nutrition and Dietetics, Harokopio University
Locations (1):
- Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared to investigators for the purpose of individual participant data meta-analysis, provided that the proposed use of the data has been approved by the Study Principal Investigator. Proposals should be directed to antonop@hua.gr. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Antonopoulou S, Fragopoulou E, Karantonis HC, Mitsou E, Sitara M, Rementzis J, Mourelatos A, Ginis A, Phenekos C. Effect of traditional Greek Mediterranean meals on platelet aggregation in normal subjects and in patients with type 2 diabetes mellitus. J Med Food. 2006 Fall;9(3):356-62. doi: 10.1089/jmf.2006.9.356. PMID 17004898
- [Background] Karantonis HC, Fragopoulou E, Antonopoulou S, Rementzis J, Phenekos C, Demopoulos CA. Effect of fast-food Mediterranean-type diet on type 2 diabetics and healthy human subjects' platelet aggregation. Diabetes Res Clin Pract. 2006 Apr;72(1):33-41. doi: 10.1016/j.diabres.2005.09.003. Epub 2005 Oct 19. PMID 16236380